CLINICAL TRIAL: NCT01562418
Title: Multi Dimensional System for Evaluating a Preventive Program for Upper Extremity Disorders Among Computer Operators
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 757-2008-IDF-CTIL
Record Dates: First submitted 2011-07-14; First posted 2012-03-23 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Musculoskeletal Disorders; Upper Extremity Pain Chronic
Keywords: Ergonomics; musculoskeletal symptoms; kinematics
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ergonomic consulting (Experimental): Ergonomic consulting without biofeedback
  Interventions: Behavioral: Standard ergonomic intervention
- Ergonomic consulting with biofeedback (Experimental): Ergonomic intervention with biofeedback
  Interventions: Behavioral: Ergonomic intervention
- general instructions (No Intervention): general instructions with no intervention
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: Ergonomic intervention — Ergonomic intervention, how to sit and work, an d muscle re education with a SurfaceElrctromyograph Biofeedback (SEMG biofeedback)
  Other Names: intervention no.2
  Arms: Ergonomic consulting with biofeedback
Behavioral: Standard ergonomic intervention — Standard ergonomic intervention , how to sit and work with computers
  Other Names: intervention no 1
  Arms: Ergonomic consulting
Behavioral: control group — general instructions no intervention
  Other Names: intervention 3
  Arms: general instructions

SUMMARY:
Computer settings points to a number of risk factors which may induce the development of Work related MSD (WRMSD). In light of the expanded use of computers and the increased occurrence of Upper Extremity (UE) WRMSD among computer operators various intervention programs have been developed and tested. Nevertheless, many of these programs do not meet the criteria of quality and level of evidence.

The main objective of this study is to use simultaneously a three dimensional (3D) kinematic analysis system, surface electromyography (SEMG) and fingertip force measurement system (Flexiforce) while typing, to test the efficacy of primary and secondary preventive intervention programs aimed at reducing MSD among computer operators.

Work hypothesis: Significant score differences will be found on the evaluation parameters between the research group which underwent ergonomic training with biofeedback, the group without feedback, and the control group.The evaluated parameters will correlate with the appearance of MSD symptoms and pain and will affect level of function.

The study will include 66 participants, programmers and computer engineers. The participants will be assigned randomly to one of three groups: 1) participants will receive ergonomic training with biofeedback; 2) participants will receive ergonomic training without biofeedback; and 3) control group, without intervention. Each group will consist of 22 participants.

Treatment efficacy will be tested both at work and in the motion lab. In the lab, 3D kinematic measurements and fingertip forces relevant to typing while entering a standard text will be measured. At the work site, anthropometric and measurements, work station measurements, posture observation and questionnaires about, psychosocial status, function and pain level will be filled The preventive program will be performed at the workstation after the preliminary data collection phase. The program will consist of one group meeting at the workplace for all employees participating in the study, and individual instruction at the workstation, including 3-6 meetings for the two research groups. Data will be collected before and after the intervention program.

ELIGIBILITY:
Inclusion Criteria:

* subjects working more than four hours per day in front of a computer and are right-hand dominant.
* Healthy or suffering from diagnoses of UE-MSD. (e.g. Rotator cuff syndrome , Lateral epicondylitis, Cubital tunnel syndrome, Carpal tunnel syndrome, Flexor-extensor peri-tendinitis or teno-synovitis of the forearm-wrist region, De Quervain's disease and Nonspecific MSD

Exclusion Criteria:

* Participants suffering from orthopedic injury or neurological deficit (with the exception of the diagnosis mentioned above).
* Medical conditions that cause swelling of the joints or hand numbness (pregnancy, diabetes, heart condition, arthritis).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-03 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal disorders measurement (MSD score) | Minimum 10 weeks and maximum 15 weeks between the first measurement and the last one.
  The MSD score of the whole body will be collected out of a self administrated questionnaire in the first meeting before intervention and in the last meeting. the score indicates the number of painful body regions that were harmful in the last week before answering the Questionnaire. Negative differences between post and pre intervention will indicate improvement in pain.

SECONDARY OUTCOMES:
Rapid Upper Limb Assessment (RULA)score | Minimum 10 weeks and maximum 15 weeks between the first measurement and the last one
  The RULA is an observation that assess the posture at work. The assessment will be held in the work place in the first meeting before intervention and in the last meeting. The score ranged between 0-7, higher score indicates higher risk for MSD. Negative differences between post and pre intervention will indicate improvement in posture at work.
Kinematic Data [range of motion ( R.O.M) and angular velocity]measured by 3D motion analysis system. | Minimum 10 weeks and maximum 15 weeks between the first measurement and the last one.
  The Kinematics of the upper extremity (fingers, wrist and elbow) will be measured in the second and in the last meeting at the motion laboratory. The second meeting will be not more than 2 weeks after the first meeting.R.O.M will be measured in degrees and the angular velocity will be presented in degrees per seconds. .Negative differences between post and pre intervention indicates improvement in R.O.M and angular velocity.
Muscle activity | Minimum 10 weeks and maximum 15 weeks between the first measurement and the last one.
  The muscle activity amplitude of the wrist and finger extensors and the upper trapezius will be measured and collected in the second meeting at the motion laboratory simultaneously with the kinematic data.The muscle amplitude will be presented as percentile of the Maximal Voluntary Contraction (MVC) of the same muscles. Higher percentage of muscle activity will indicate higher muscle load. Negative differences between post and pre intervention indicates improvement in muscle activity.
Psychosocial job characteristics assessment (DCSQ) | Minimum 10 weeks and maximum 15 weeks between the first measurement and the last one.
  The D.C.S.Q will be measured by a self administrated questionnaire in the first meeting before intervention and in the last meeting. The job demands score range between 5-25 and the decision latitude score range between 8-40. Low level of job demands and high decision latitude indicates low level of stress at work.

CONTACTS AND LOCATIONS:
Overall Officials: Yafi Levanon, MsC, Study Director — Sheba Medical Center , Tel aviv University
Locations (1):
- Motion Laboratory, Sheba medical center, Ramat Gan, Israel